CLINICAL TRIAL: NCT05098314
Title: Impact of Personalized Interventions to Raise Teleconsultation Awareness: The Case of the Cicat-Occitanie Network and Healthcare Professionals in Lozère's EHPADs
Brief Title: Impact of Personalized Interventions to Raise Teleconsultation Awareness in EHPAD
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0373
Record Dates: First submitted 2021-10-18; First posted 2021-10-28 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Wound Healing Disorder
Keywords: telemedicine; Cluster Randomised Trial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EHPAD with personalized interventions: EHPAD with personalized interventions.
  Interventions: Other: Personalized interventions regarding the Cicat-Occitanie network
- EHPAD without personalized interventions: EHPAD without personalized interventions

INTERVENTIONS:
Other: Personalized interventions regarding the Cicat-Occitanie network — First of all, healthcare professionals from EHPAD in the intervention arm were invited by email to answer a closed questionnaire. It was built by the authors, on Google forms, and consisted of 11 questions divided into 2 sections.
  Section 1 collected data about the participants. In section 2, they were asked to score from 0 to 4 (ranging from "not at all "to" a lot ") the various obstacles to teleconsultations reported by the literature.
  Groups: EHPAD with personalized interventions

SUMMARY:
The cicat-occitanie network offers expertise for health professionals concerning wound care, in particular through teleconsultations. This study aimed to understand the obstacles reported by healthcare professionals in Lozere's EHPAD related to the use of this network. This cluster randomized controlled trial also sought to evaluate the effect of personalized intervention for each EHPAD on the use of this network.

ELIGIBILITY:
Inclusion criteria:

- Be a resident in Lozère's EHPAD

Exclusion Criteria:

- Patient who reject the study protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All residents of Lozère's EHPADs
Sampling Method: Probability Sample
Enrollment: 1612 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-09-17 (Actual)

PRIMARY OUTCOMES:
Requests rate for teleconsultations | 3 months
  Requests rate for teleconsultations with the Cicat-Occitanie network by Lozère's EHAPDs.
  Incidence in resident-year of new requests of teleconsultations from the Cicat-Occitanie network by health professionals from Lozère's EHPADs. Calculated via numbers transmitted by the Cicat-Occitanie network 3 months after the intervention and the number of residents in each EHPAD.

SECONDARY OUTCOMES:
Human obstacles linked to the use of teleconsultations | 4 months
  Human obstacles linked to the use of teleconsultations with the Cicat-Occitanie network reported by health professionals in Lozère's EHPAD Rating of the different human obstacles from 0 to 4 (not at all to a lot) by the health professionals in EHPAD of Lozère. This was collected through an online questionnaire.
Organizational obstacles linked to the use of teleconsultations | 4 months
  Organizational obstacles linked to the use of teleconsultations from the Cicat-Occitanie network reported by health professionals in Lozère's EHPAD.
  Rating of the different organizational obstacles from 0 to 4 (not at all to a lot) by the health professionals in EHPAD of Lozère. This was collected through an online questionnaire.
Economic obstacles linked to the use of teleconsultations | 4 months
  Economic obstacles linked to the use of teleconsultations from the Cicat-Occitanie network reported by health professionals in Lozère's EHPAD.
  Rating of the different obstacles from 0 to 4 (not at all to a lot) by the health professionals in EHPAD of Lozère. This was collected through an online questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Bastien Paul, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC